CLINICAL TRIAL: NCT00403533
Title: Assessment of the Antiviral Effect of Atorvastatin on Hepatitis C Virus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-P-000138/1; AASLD advanced hepato. grant
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Last update posted 2006-11-23 (Estimated); Status verified 2006-11

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; viral load; antiviral therapy; cholesterol; atorvastatin
MeSH Terms: conditions — Hepatitis C

INTERVENTIONS:
Drug: 20 mg of atorvastatin daily

SUMMARY:
We hypothesize that atorvastatin will decrease HCV viral load in patients taking the medication.

Cholesterol is needed for HCV virion production. Cell culture studies have shown that atorvastatin (an HMG-CoA reductase inhibitor) decreases HCV viral replication. As atorvastatin has been proven to decrease heart attack and stroke in patients with high cholesterol, this medication is indicated for the treatment of elevated cholesterol in at risk individuals. Therefore we propose to study the effect atorvastatin has on the viral load of patients initiated on atorvastatin therapy for their elevated cholesterol.

DETAILED DESCRIPTION:
Men and women ages 30 to 80 infected with HCV viremia whose physician has determined need cholesterol lowering medication will be recruited by the study investigators from Massachusetts General Hospital.

The study investigators will approach the potential subject after the referring doctor has ascertained that the potential subject is interested in meeting with the investigator.

Each subject who consents will undergo phlebotomy of 10 cc of blood three times. Once prior to the initiation of atorvastatin to measure the patients viral load. In addition, patients will undergo phlebotomy 4 and 12 weeks after the initiation of atorvastatin. The week 12 phlebotomy is required in all patients started on atorvastatin to monitor for side effects. Therefore patients who enroll in this study will undergo one additional phlebotomy. As part of our study an extra 10 cc of blood will be taken at these times to measure the patients HCV viral load.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic HCV.
* Patients who need treatment for their elevated cholesterol:

  * Total cholesterol >240 or
  * LDL >160 without cardiac risk factors or
  * LDL >130 with two cardiac risk factors (hypertension, smoker, family history of heart attach, or HDL <40 for men or <50 for women) or
  * LDL >100 with diabetes or known coronary artery disease

Exclusion Criteria:

* Impaired mental ability preventing a subject from understanding the protocol or from completing the entire study.
* HCC
* A history of an adverse reaction to any HMG CoA reductase inhibitor.
* Patients who are on HCV treatment, who plan to initiate HCV treatment within 3 months, or who discontinued HCV treatment within the last 3 months.
* Patients whose aminotransferases are > 5 times the upper limit of normal.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2006-02; Study Completion 2006-07

PRIMARY OUTCOMES:
Paired comparison of pretreatment viral load to post-treatment 12 week viral load

SECONDARY OUTCOMES:
Paired comparison of pretreatment viral load to post-treatment 4 week viral load

CONTACTS AND LOCATIONS:
Overall Officials: Raymond T Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ikeda M, Abe K, Yamada M, Dansako H, Naka K, Kato N. Different anti-HCV profiles of statins and their potential for combination therapy with interferon. Hepatology. 2006 Jul;44(1):117-25. doi: 10.1002/hep.21232. PMID 16799963
- [Background] Kapadia SB, Chisari FV. Hepatitis C virus RNA replication is regulated by host geranylgeranylation and fatty acids. Proc Natl Acad Sci U S A. 2005 Feb 15;102(7):2561-6. doi: 10.1073/pnas.0409834102. Epub 2005 Feb 7. PMID 15699349
- [Background] Aizaki H, Lee KJ, Sung VM, Ishiko H, Lai MM. Characterization of the hepatitis C virus RNA replication complex associated with lipid rafts. Virology. 2004 Jul 1;324(2):450-61. doi: 10.1016/j.virol.2004.03.034. PMID 15207630